CLINICAL TRIAL: NCT04423263
Title: Perioperative Prophylactic Bilateral Internal Iliac Artery Occlusion in Placenta Accreta: a Randomized Trial
Brief Title: Internal Iliac Artery Occlusion in Placenta Accreta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Voon Hian Yan (Other)
Responsible Party: Sponsor-Investigator, Voon Hian Yan, Consultant Maternal Fetal Medicine Specialist, Sarawak General Hospital
Organization: Sarawak General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Research ID 55302
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Placenta Accreta
Keywords: balloon occlusion; iliac artery; interventional radiology; postpartum hemorrhage; blood transfusion
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Receives bilateral internal iliac artery occlusion
  Interventions: Procedure: Bilateral internal iliac artery balloon occlusion
- Control (Active Comparator): Does not receive bilateral internal iliac artery occlusion
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Bilateral internal iliac artery balloon occlusion — Bilateral internal iliac artery balloon placement under fluoroscopic guidance preoperatively which will be occluded intraoperatively based on existing local protocol
  Arms: Intervention
Procedure: Control — Surgical approach similar to intervention arm, except bilateral internal iliac artery occlusion
  Arms: Control

SUMMARY:
This is a randomized study to assess the efficacy of prophylactic bilateral internal iliac artery occlusion performed prior to planned surgical management for placenta accreta spectrum (PAS). The intervention group would receive balloon occlusion, ureteric stenting and caesaeran hysterectomy while the control group would undergo the same procedure, excluding balloon occlusion. The primary outcome is to demonstrate a three pint or greater reduction in pack cell transfusion requirement.

DETAILED DESCRIPTION:
Interventional radiology, including internal iliac artery occlusion, has been used as an adjunct in the management of placenta accreta spectrum (PAS). Retrospective studies have shown benefit in terms of reduction of blood loss. However, studies reported in literature vary widely in terms of the exact surgical procedure undertaken, in conjunction with the radiological intervention. The radiological intervention itself lacks standardization, occurring at different anatomical levels, ranging from infrarenal aortic occlusion to internal iliac or uterine artery. Furthermore, there have been reported cases of arterial thrombosis associated with arterial occlusion.

We sought to clarify the effectiveness of a standardized approach , where perioperative bilateral internal iliac artery occlusion is performed followed by bilateral ureteric stenting and caesarean hysterectomy. The control group would undergo the exact procedure, excluding internal iliac artery occlusion. Patients would be randomized but neither the patient nor surgeon could be blinded.

The primary outcome would be to demonstrate a three pint or greater reduction in packed cell transfusion. Secondary outcomes include a difference in estimated blood loss, additional blood product transfusion, unplanned additional surgical procedure, serious complications arising from internal iliac artery occlusion, total procedural time and early neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with prenatally diagnosed placenta accreta spectrum

Exclusion Criteria:

* Women who declined to participate
* Women with bleeding diathesis or severe thrombocytopenia <100k x 1,000,000/L
* Surgery performed prior to 28 weeks of gestation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pack cell transfusion | First 7 days post-operatively
  To detect a three pint reduction in pack cell transfusion

SECONDARY OUTCOMES:
Other blood components | First 7 days post-operatively
  Platelets, fresh fozen plasma, cryoprecipitate
Unplanned perioperative surgical procedures | First 7 days post-operatively
  Internal iliac artery ligation, abdominal packing, relaparotomy
Complication from internal iliac occlusion | First 14 days post-operatively
  death, arterial thrombosis, aneurysm, hematoma requiring evacuation

OTHER OUTCOMES:
Operative time | Perioperative
  Total time taken for procedure
Neonatal complication | First 24 hours
  Apgar, cord pH, resuscitation, neonatal intensive care admission

CONTACTS AND LOCATIONS:
Overall Officials: Hian Yan Voon, MRCOG, Principal Investigator — Sarawak General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and anonymized information including demographics, primary and secondary outcomes
Supporting Information: Study Protocol
Time Frame: 36 months from the date of completion of study
Access Criteria: Written permission to authors and submission of complete protocol

REFERENCES:
- [Background] Chen M, Liu X, You Y, Wang X, Li T, Luo H, Qu H, Xu L. Internal Iliac Artery Balloon Occlusion for Placenta Previa and Suspected Placenta Accreta: A Randomized Controlled Trial. Obstet Gynecol. 2020 May;135(5):1112-1119. doi: 10.1097/AOG.0000000000003792. PMID 32282608
- [Background] Salim R, Chulski A, Romano S, Garmi G, Rudin M, Shalev E. Precesarean Prophylactic Balloon Catheters for Suspected Placenta Accreta: A Randomized Controlled Trial. Obstet Gynecol. 2015 Nov;126(5):1022-1028. doi: 10.1097/AOG.0000000000001113. PMID 26444128